CLINICAL TRIAL: NCT05352893
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Adult Subjects With Generalized Pustular Psoriasis
Brief Title: Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Subjects With GPP
Acronym: GEMINI1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB019-301
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2023-09

CONDITIONS: Generalized Pustular Psoriasis
Keywords: IL-36 Receptor; Interleukin 36; Imsidolimab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On Day 1, eligible subjects will be randomized in a 1:1:1 ratio to receive a single intravenous (IV) high dose imsidolimab, low dose imsidolimab, or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IV high dose Imsidolimab, other name ANB019 (Experimental): ANB019 Biological Humanized Monoclonal Antibody High Dose
  Interventions: Drug: Imsidolimab high dose
- IV low dose Imsidolimab, other name ANB019 (Experimental): ANB019 Biological Humanized Monoclonal Antibody Low Dose
  Interventions: Drug: Imsidolimab low dose
- IV Placebo (Placebo Comparator): Placebo Solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Imsidolimab high dose — intravenous
  Other Names: ANB019
  Arms: IV high dose Imsidolimab, other name ANB019
Drug: Imsidolimab low dose — intravenous
  Other Names: ANB019
  Arms: IV low dose Imsidolimab, other name ANB019
Other: Placebo — intravenous
  Arms: IV Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of imsidolimab compared with placebo in adult subjects with generalized pustular psoriasis (GPP).

DETAILED DESCRIPTION:
This study will also characterize the pharmacokinetic (PK) profile of imsidolimab and explore the immunogenicity of imsidolimab in subjects with GPP.

ELIGIBILITY:
Inclusion Criteria:

-Subject has a BSA affected with pustules (excluding palms and soles) ≥ 5%, a GPPPGA score ≥ 3 (moderate severity), and a PRS score ≥ 3 (moderate severity) at Day 1

Exclusion Criteria:

* Subject has other form of psoriasis excluding psoriasis vulgaris
* Subject flare is so severe that patient's life is at risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving Generalized Pustular Psoriasis Physician's Global Assessment (GPPPGA) score of 0 (clear) or 1 (almost clear) | week 4
  Baseline to 0 (clear) or 1 (almost clear)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (5):
  - Site 109, Largo, Florida
  - Site 105, Louisville, Kentucky
  - Site 101, Ann Arbor, Michigan
  - Site 108, Dallas, Texas
  - Site 102, Springville, Utah
- Australia (2):
  - Site 35-101, Melbourne
  - Site 35102, Sydney
- Georgia (5):
  - Site 59104, Batumi
  - Site 50103, Tbilisi
  - Site 59-101, Tbilisi
  - Site 59-105, Tbilisi
  - Site 59102, Tbilisi
- Germany (4):
  - Site 17102, Bensheim
  - Site 17104, Bonn
  - Site 17103, Hanau
  - Site 17105, Würzburg
- Malaysia (6):
  - Site 42104, Cheras
  - Site 42106, Johor Bahru
  - Site 42105, Kota Bharu
  - Site 42101, Kuala Lumpur
  - Site 42102, Muar town
  - Site 42103, Putrajaya
- Morocco (3):
  - Site 64-102, Casablanca
  - Site 64-103, Casablanca
  - Site 64-101, Oujda
- Poland (5):
  - Site 30104, Krakow
  - Site 30105, Lodz
  - Site 30103, Ossy
  - Site 30101, Rzeszów
  - Site 30102, Wroclaw
- Romania (3):
  - Site 31-102, Bucharest
  - 31-101, Cluj-Napoca
  - Site 31-103, Iași
- Site 38-101, Svidník, Slovakia
- South Korea (4):
  - Site 45101, Pusan
  - Site 45102, Seoul
  - Site 45103, Seoul
  - Site 45104, Seoul
- Spain (5):
  - Site 24-101, Barcelona
  - Site 24-104, Las Palmas de Gran Canaria
  - Site 24-102, Madrid
  - Site 24-103, Madrid
  - Sie 24-105, Valencia
- Taiwan (4):
  - Site 63101, Kaohsiung City
  - Site 63102, Taipei
  - Site 63103, Taipei
  - Site 64104, Taipei
- Thailand (4):
  - Site 46101, Bangkok
  - Site 46102, Chiang Mai
  - Site 46104, Khon Kaen
  - Site 46103, Pathum Thani
- Tunisia (3):
  - Site 62-101, Sfax
  - Site 62-102, Sousse
  - Site 62-103, Tunis
- Turkey (Türkiye) (6):
  - Site 33-102, Ankara
  - Site 33-103, Antalya
  - Site 33-105, Istanbul
  - Site 33-106, Istanbul
  - Site 33-107, Istanbul
  - Site 33-104, Nilufer

IPD SHARING:
Plan to Share IPD: No